CLINICAL TRIAL: NCT06314945
Title: Diagnostic Value of Recto-perineal Ultrasound in Perianal Fistula; Pre Versus Intraoperative Findings: a Comparative Cross Section Study
Brief Title: Diagnostic Value of Recto-perineal Ultrasound in Perianal Fistula
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, Principal Investigator, Zagazig University
Other Study IDs: #11280-4\12-2023
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Perianal Fistula
Keywords: recto-perineal ultrasound; perianal fistula; trans-sphincteric

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perianal fistula is a common anal problem. It needs only surgery. MRI is the best preoperative diagnostic tool, but it is demanding as it is expensive, time consuming and needs an experienced radiologist. So, we tried to find an alternative diagnostic tool which is cheaper, time saving and accurate and comparing its preoperative reports with intraoperative findings.

study was held in surgery department in Zagazig University Hospitals from September 2023 to March 2024. It included 93 patients with perianal fistula who were diagnosed clinically and radiological by trans recto-perineal ultrasound and comparing pre-operative ultrasound findings with intra-operative surgical findings.

ELIGIBILITY:
Inclusion Criteria:

* Perianal abscess and\or fistula
* Patients who accidently discovered during transvaginal ultrasound.
* Age group between above 18 years old

Exclusion Criteria:

* Informed consent refusal.
* Proved anal malignancy.
* Patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: only patients with perianal fistula or abscess in zagazig university hospitals who admitted during the study duration were included in the study
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
age | from 2 to 3 days before operation
  age of patient was recorded in years
sex | from 2 to 3 days before surgery
  sex of patients was recorded as male or female
body mass index | from 2 to 3 days before surgery
  patient BMI was recorded by dividing weight in kg by length square in meters
history of abscess drainage | from 2 to 3 days before surgery
  history of perianal abscess was recorded
Internal opening | from 2 to 3 days pre-operative and intraoperatively
  presence and site of internal opening was assessed by digital rectal examination and utrasound
fistula branches | from 2 to 3 days pre-operative and intraoperatively
  presence of fistula branches and their number were assessed by ultrasound and during surgery
type fistulous tract | from 2 to 3 days pre-operative and intraoperatively
  type of fistula was detected in relation to anal sphincters by ultrasound and intraoperative
abscess cavity | from 2 to 3 days pre-operative and intraoperatively
  presence or absence of abscess cavity was assessed in ultrasound and intraoperative

SECONDARY OUTCOMES:
other anal disease | from 2 to 3 days before surgery
  presence or absence of other anal disease like anal fissure, piles or inflammatory bowel disease from medical records of the patients
external openings | from 2 to 3 days pre-operative and intraoperatively
  number and site of external openings was assessed by clinical and radiological examination
anal discharge | from 2 to 3 days before surgery
  presence or absence of anal discharge, its color, odor and viscosity were assessed by history of soiling underwear and clinical examination by soiling of gloves or direct vision of discharge during digital rectal examination

CONTACTS AND LOCATIONS:
Overall Officials: Reham Zakaria, PhD, Principal Investigator — faculty of medicine Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt